CLINICAL TRIAL: NCT04249063
Title: FUndal Block During NovaSure enDometrial AbLation to Reduce Intraoperative PAIN: A Randomized Controlled Trial
Brief Title: Fundal Block in Pre-menopausal Women to Reduce Pain During Outpatient-based Endometrial Ablation (FUNDAL-PAIN)
Acronym: FUNDAL-PAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Principal Investigator, Darrien Rattray, Principal Investigator, Clinical Associate Professor, Department of Obstetrics and Gynecology, Saskatchewan Health Authority - Regina Area
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SaskHealthAuthority
Record Dates: First submitted 2020-01-26; First posted 2020-01-30 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pain
Keywords: Abnormal Uterine Bleeding; Endometrial Ablation; NovaSure; Pain
MeSH Terms: conditions — Pain; Metrorrhagia | interventions — Lidocaine; Saline Solution; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient (participant), physician (care provider), recovery nurse (outcomes assessor) and researcher team (investigator) will all be blinded to the intervention. Only the assisting nurse dedicated to procedural setup will be aware of the allocated intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): NovaSure EA with an injection of local anaesthetic into the fundus. Paracervical block and procedural sedation as per usual.
  Interventions: Drug: Xylocaine 1 % and Normal Saline
- Control Group (Placebo Comparator): NovaSure EA with an injection of normal saline into the fundus. Paracervical block and procedural sedation as per usual.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Xylocaine 1 % and Normal Saline — 3cc aliquots of local anaesthetic will be injected into the right and left cornual regions and centrally in the fundus. This will be achieved by using a flexible hysteroscopic needle.
  Other Names: Local anaesthetic
  Arms: Treatment Group
Drug: Normal Saline — 3cc aliquots of normal saline will be injected into the right and left cornual regions and centrally in the fundus. This will be achieved by using a flexible hysteroscopic needle.
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
The objective of this study is to assess the efficacy of a fundal block in reducing women's perception of pain during NovaSure endometrial ablation (EA) in an outpatient-based setting.

DETAILED DESCRIPTION:
The researchers aim to determine whether participants receiving the paracervical and fundal block (experimental group) achieve clinically and statistically significant reductions in self-reported pain during NovaSure EA, as compared to those receiving paracervical block (control group). All women will obtain concurrent procedural sedation. Women's perception of pain will be recorded on a scale from 0 to 10 using the visual analogue scale (VAS).

The researchers hypothesize that the participants receiving combined paracervical and fundal block will experience less pain during the active procedure, as compared to those receiving paracervical block alone.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal uterine bleeding
* Pre-menopausal as determined by the presence of menstrual cycles
* Must have completed their family or have no desire to preserve fertility
* Uterus and cervix must meet eligibility criteria; based on hysteroscopy exam performed by the physician prior to the ablation procedure
* Must be a female participant 25-55 years of age

Exclusion Criteria:

* Any uterine characteristics that preclude performing EA
* Past allergic reactions to local anaesthetic
* Weight <50kg
* Submucous fibroids requiring myomectomy
* Lack of patient consent

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 288 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative pain | 30 seconds into active ablation procedure
  Thirty seconds into the active NovaSure EA procedure, all participants will be asked the same standardized question to rate their pain. The question will be posed by the registered nurse assisting the physician, and the women will score their perception of pain on a scale from 0 to 10 using the VAS.

SECONDARY OUTCOMES:
Post-operative pain | 1 hour post-procedure
  Using the VAS, all participants will be asked to rate their pain 1 hour post-procedure.
Rescue analgesics/and or sedation | From time of active ablation procedure to discharge from unit (t = 0 sec to t = ~3hrs).
  The use of additional rescue analgesics/and or sedation during the active ablation procedure and post-operative period will be recorded and compared between groups.
Adverse reactions | From time of active ablation to discharge from unit ( t= 0 sec to t = ~3hrs).
  Any adverse reactions that occur in response to the fundal injections during and following the procedure will be recorded and compared between groups.
Acceptability of the procedure | Post-procedure prior to discharge (t = ~3hrs).
  The acceptability of the ablation procedure will be evaluated between groups by asking each participant if they would recommend the procedure to a friend.

CONTACTS AND LOCATIONS:
Overall Officials: Darrien Rattray, MD, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Gynaecology & Pediatric Associates, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No